CLINICAL TRIAL: NCT01259739
Title: The Impact of Dietary Cocoa Flavanols on Cardio-pulmonary Exercise Capacity in Human.
Brief Title: Cocoa Flavanols and Exercise Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Tienush Rassaf, MD, PhD, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Flavanols - Exercise
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Exercise Capacity
Keywords: trained cyclists; no medications; no diseases; non-smokers
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavanol rich cocoa (Experimental): (596 mg), dissolved in water, twice daily intervention
  Interventions: Other: Cocoa
- flavanol poor cocoa drink (Experimental): ( 13mg) dissolved in water, twice daily intervention
  Interventions: Other: Cocoa

INTERVENTIONS:
Other: Cocoa — dissolved in water twice-daily intervention

SUMMARY:
The purpose of this study is to characterize the potential improvement of cocoa flavanols on exercise capacity in highly trained cyclist. A placebo-controlled double-blinded randomized control study will be performed in 13 highly trained cyclist (crossover design). Participants will perform a baseline exercise testing on an ergometer. They will receive either a flavanol-poor or flavanol rich cocoa drink twice daily for one week before a second and third exercise testing is performed. The order of drinks is randomized and balanced (high-flavanol-->low-flavanol drink or low-flavanol drink-->high-flavanol drink)

DETAILED DESCRIPTION:
13 participants (highly-trained cyclist, accustomed to exercise testing on ergometers will be enrolled (VO2max>50 ml/kg, FMD >5%, non-smokers, no medication, no diseases, age 20-36, male).

Baseline Testing:

Participants will perform a baseline testing consisting of an ergometric test with a step-wise increase of workload until exhaustion to determine lactate anaerobic threshold and cardio-pulmonary exercise capacity. Vascular function is monitored by Doppler Ultrasound.

In a second test, participants will perform a time trial (goal: as fast as possible)

Flavanol intervention Participants will twice daily receive either a flavanol-poor cocoa drink (13mg/dl)or a flavanol-rich cocoa drink (596mg/dl) over a period of 7 days. Order is randomized and balanced. Subjects will crossover to the second arm after a washout period of 7 days.

Testing performed on baseline day is repeated after the intake of both drinks

In a subgroup of n=6 participants, we will test whether the blood pressure cuff maneuver used for FMD will itself modify nitrite levels. For this the manuever will be completed 4 times and compared to n=6 untreated controls. in another subgroup 6 participants will receive 4times the maneuver but reperfusion will be limited by means of an ultrasound probe.

ELIGIBILITY:
Inclusion Criteria:

* highly trained cyclists (VO2 peak > 50 ml/kg bodyweight)
* refrain from cocoa ingestion during trial
* training continued throughout testing
* > 20 years
* male

Exclusion Criteria:

* > 36 years
* poor endothelial function
* acute infection
* any chronic heart or pulmonary disease
* arrhythmias
* acute or chronic renal failure
* smokers
* cardio-vascular risk factors : diabetes mellitus, hypertension, hyperlipidemia
* intake of nutrition supplements (l-arginine, creatinine)
* intake of WADA listed doping substances

Ages: 20 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary exercise capacity (time to complete time trail, lactate anaerobic threshold, cardio-pulmonary exercise capacity | 7 days

SECONDARY OUTCOMES:
Endothelial function | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, PhD, Principal Investigator — Heinrich Heine University Düsseldorf, NRW, Germany; Malte Kelm, MD, PhD, Study Chair — Heinrich Heine University Düsseldorf, NRW, Germany
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Rassaf T, Totzeck M, Hendgen-Cotta UB, Shiva S, Heusch G, Kelm M. Circulating nitrite contributes to cardioprotection by remote ischemic preconditioning. Circ Res. 2014 May 9;114(10):1601-10. doi: 10.1161/CIRCRESAHA.114.303822. Epub 2014 Mar 18. PMID 24643960
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie